CLINICAL TRIAL: NCT04362865
Title: Investigation of the B- and T-cell Repertoire and Immune Response in Patients With Acute and Resolved COVID-19 Infection
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 200103; 20-C-0103
Record Dates: First submitted 2020-04-24; First posted 2020-04-27 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: COVID-19
Keywords: Pandemic; Coronavirus; SARS-CoV-2; Natural History
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 infection: Patients with confirmed or suspected COVID-19 infections
- No COVID-19 infection: Patients without confirmed or suspected COVID-19 infections (i.e., normal donors)

SUMMARY:
Background:

People who get infected with COVID-19 have an unpredictable risk to worsen and die. This makes it hard to decide who can quarantine at home and who should be treated at a hospital. Researchers think the risk may be related to how a person s B and T cells respond to the virus. B and T cells are the major components of a person s immune response. B and T cells responding to the virus with a favorable pattern may lead to recovery, and this favorable pattern may be helpful to establish. If people in a vaccine trial get this same favorable pattern when responding to a vaccine, this may be a useful early signal that the vaccine will be successful.

Objective:

To examine how immune cells respond to COVID-19 infection.

Eligibility:

Adults ages 18 and older who have a confirmed or suspected COVID-19 infection or had COVID-19 in the past.

Also, healthy donors with no suspected COVID-19 infection

Design:

Participants will be screened with medical record review.

Participants will be tested with a research assay to determine who was infected with COVID-19 and who was not. This test will be used to understand research results, not to advise patients.

Participants with active infection must be isolated, usually in a hospital.

Other participants may give blood samples at NIH or at their local doctor s office or lab.

Participants may give blood samples up to three times a week for a total of ten times, and may also give blood samples after starting a vaccine trial.

Participants will be contacted by phone or email every 2 months for up to 2 years.

DETAILED DESCRIPTION:
Background:

Patients infected with COVID-19 have an unpredictable risk to worsen and die, making it difficult to decide who can quarantine at home and who should be monitored for respiratory failure as an inpatient. This risk may be related in part to the patient s immune response which can be characterized with respect to the B- and T-cell repertoire. Determining patterns of immune response which correlate with clinically effective immunity may help in determining risk.

Patients receiving a vaccine for COVID-19 are tested for antibody production, but ultimately protection from infection and survival are the most important endpoints, which will take time. If patients can be checked for a pre-defined favorable pattern of immune response, it may significantly speed selection of effective candidate vaccines.

In patients with hematologic malignancies, including patients with hairy cell leukemia (HCL) who we have extensive experience treating, we do not know if we should be steering away more from treatments which harm B-cell immunity, like rituximab or obinutuzumab, or steering away more from treatments which harm T-cell immunity, like purine analogs. Characterizing the immune response in COVID-19 patients will quickly answer this question.

Objective:

To characterize immune response in patients with current or prior COVID-19 infection

Eligibility:

Age 18 years or older

Patients with known or suspected COVID-19 infection, or normal donors (i.e., those individuals without COVID-19)

Design:

Blood samples will be collected for research to characterize immune response.

In individuals with suspected or known current or prior COVID-19, samples will be obtained up to every three days but no more than 10 times overall during the acute phase of infection. After recovery, samples will be collected up to ten times overall. In individuals without COVID-19 at the time of enrollment (i.e., normal donors), samples will be collected at least once; in the case of future COVID-19 infection, samples may be collected at the same times during/post-infection as an individual with COVID-19 at enrollment.

Additional blood and urine samples may be collected in all subjects before and after the receipt of COVID-19-related vaccination.

All subjects will be followed for approximately 2 years.

This protocol does not involve treatment. The accrual ceiling is set at 745 subjects.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Individuals who meet one of the following groups:

  * Patients with a confirmed or suspected diagnosis of COVID-19 infection, current or resolved; or,
  * Normal donors. Note: For the purpose of this study, normal donors are those without a known current, past, or suspected COVID-19 infection; individuals may have other medical comorbidities or conditions.
* At least 18 years of age
* Ability of patient or Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent document

EXCLUSION CRITERIA: Individuals with COVID-19

- Desire of the patient or normal donor not to submit samples, or medical contraindication to sending samples.

EXCLUSION CRITERIA: Normal Donors

- No Exclusions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary clinical
Sampling Method: Non-Probability Sample
Enrollment: 679 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
Characterize immune response | Ongoing
  characterize immune response in patients with active or prior COVID-19 infection

SECONDARY OUTCOMES:
Immune response and outcome | ongoing
  determine if there is a correlation between the pattern of immune response to COVID-19 and outcome in patients with acute or resolved infection
B- and T-cell arm immune response | ongoing
  determine if the B- or T-cell arm of the immune response is more active in responding to COVID-19 infection

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Kreitman, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (4):
- United States (4):
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Medstar Franklin Square Medical Center, Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Medstar Montgomery Medical Center, Olney, Maryland

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- [Derived] Kreitman RJ, James L, Feurtado J, Eager H, Sierra Ortiz O, Gould M, Shpilman I, Zhou H, Burbelo PD, Cohen JI, Wang HW, Yuan CM, Arons E. COVID-19 vaccination in patients with classic and variant hairy cell leukemia. Blood Neoplasia. 2024 Aug 28;1(4):100035. doi: 10.1016/j.bneo.2024.100035. eCollection 2024 Dec. PMID 40552139
- [Derived] Arons E, Henry K, Haas C, Gould M, Tsintolas J, Mauter J, Zhou H, Burbelo PD, Cohen JI, Kreitman RJ. Characterization of B-cell receptor clonality and immunoglobulin gene usage at multiple time points during active SARS-CoV-2 infection. J Med Virol. 2023 Oct;95(10):e29179. doi: 10.1002/jmv.29179. PMID 37877800
- [Derived] Kreitman RJ, Yu T, James L, Feurtado J, Eager H, Ortiz OS, Gould M, Mauter J, Zhou H, Burbelo PD, Cohen JI, Wang HW, Yuan CM, Arons E. COVID-19 in patients with classic and variant hairy cell leukemia. Blood Adv. 2023 Dec 12;7(23):7161-7168. doi: 10.1182/bloodadvances.2023011147. PMID 37729613
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-C-0103.html